CLINICAL TRIAL: NCT03901430
Title: Designing a Culturally Appropriate Group Navigation Model to Improve Mental and Emotional Health Equity for Spanish-Speaking Latina Women
Brief Title: Designing a Mental Health Model for Latina Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 18-305; U54MD004811 (NIH)
Record Dates: First submitted 2019-04-01; First posted 2019-04-03 (Actual); Results first posted 2023-02-06 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2019-04

CONDITIONS: Mental Health Wellness 1; Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Masking Description: Participants are given ID numbers and all data is coded with ID number
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Class (Experimental): Group navigation model
  Interventions: Behavioral: Group navigation model

INTERVENTIONS:
Behavioral: Group navigation model — In a series of peer group sessions facilitated by Guadalupe Fuentes, a CHW who designed the model, we will create a culturally-appropriate, non-stigmatizing group intervention. The group process will allow participants to explore their own MEH, better understand the ways that mental health influences well-being and everyday dynamics of their lives, and to develop empowering knowledge and action plans through the support of other women.

SUMMARY:
The goal of this study is to implement such an approach conceptualized by a community health worker (CHW) to pilot an innovative, multi-level intervention to address social and structural determinants that negatively influence MEH disparities for Latinas from low-income households. The proposed research integrates CHW navigation with group peer support. Both of these strategies have been shown to be culturally appropriate and effective for improving a variety of health outcomes with this population. Our transdisciplinary, community-engaged team will use a convergent parallel mixed method research design to assess the feasibility of the intervention and its impact on six domains of interest: 1) emotional support, 2) informational support, 3) depression, 4) social isolation, 5) empowerment, and 6) social determinants needs. To prepare for future extramural funding, the investigators will include development of an advocacy plan for multi-level social change impact.

DETAILED DESCRIPTION:
Hispanic women (Latinas) experience mental and emotional health (MEH) concerns and disorders that often go unrecognized by health providers, and even when recognized, Latinas have low-levels of treatment follow-through with biomedical modalities. Using a novel community-directed, solution-based approach to increase access to existing services and nurture culturally meaningful social relationships, it is possible to address social determinants of health and reduce these disparities.

The goal of this study is to implement such an approach conceptualized by a community health worker (CHW) to pilot an innovative, multi-level intervention to address social and structural determinants that negatively influence MEH disparities for Latinas from low-income households. The proposed research integrates CHW navigation with group peer support. Both of these strategies have been shown to be culturally appropriate and effective for improving a variety of health outcomes with this population. Our transdisciplinary, community-engaged team will use a convergent parallel mixed method research design to assess the feasibility of the intervention and its impact on six domains of interest: 1) emotional support, 2) informational support, 3) depression, 4) social isolation, 5) empowerment, and 6) social determinants needs. To prepare for future extramural funding, the investigators will include development of an advocacy plan for multi-level social change impact.

Aim 1. Create a group navigation model to improve mental and emotional health equity for Spanish-speaking Latina women. In a series of peer group sessions facilitated by Guadalupe Fuentes, a CHW who designed the model, the investigators will create a culturally-appropriate, non-stigmatizing group intervention. The group process will allow participants to explore their own MEH, better understand the ways that mental health influences well-being and everyday dynamics of their lives, and to develop empowering knowledge and action plans through the support of other women. The investigators will document group discussions, processes, and themes, gather information about women's explanatory models of MEH, and administer a multidimensional survey to capture information about the domains of interest. Through individual case management, Fuentes will work individually with women from the groups to identify their specific social and structural determinants needs, assist them to make an individual action plan, provide them with information about available resources, and help them navigate systems and access resources and services. The investiagtors will document participant needs and navigation outcomes. Hypotheses: Participation will decrease depression, social isolation, and social determinants needs, and increase emotional support, informational support, and women's sense of empowerment.

Aim 2. Create an advocacy plan. With data gathered in group meetings and individual navigation sessions, the investigators will identify social and structural barriers that negatively influence participants' MEH outcomes and ability to access resources and services. The investigators will create an advocacy plan to address structural and policy barriers that can be implemented by CHWs and advocacy groups in the future. Hypotheses: The investigators will be able to identify factors that negatively influence the MEH and well-being of Latinas. They hypothesize that in the future, this knowledge can be used to develop a strategic plan with the potential to address socio-structural and policy barriers through advocacy.

Aim 3. Assess the feasibility of the intervention. The investigators will track recruitment, attrition, attendance at group sessions, and attendance at individual CHW navigation meetings.The investigators will gather survey data and qualitative data to document participant experiences with and perceptions of the group process, working with the CHW, and the value of the intervention. Hypotheses: The intervention pilot will be feasible, acceptable, valuable, and culturally appropriate.

Expected Outcome. This pilot study will use team science to test an intervention that emerged organically in the community and contribute to building the next generation of health disparities research using knowledge generated through solution-based investigation as the foundation for submitting an NIH R21 research proposal.

ELIGIBILITY:
Inclusion Criteria:

* female over 18 Spanish-speaking economically disadvantaged

Exclusion Criteria:

* male under 18 non-Spanish-speaking non-economically disadvantaged

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 21 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-03-18 (Actual); Study Completion 2020-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Cacari Stone, Ph.D., Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: During month #2 prior to the start of the intervention, Fuentes recruited 30 participants through the Pathways Program, the Simplemente Salud Clinic and Centro Sávila. In the course of regular meetings with clients who request a range of services, she will identify and invite those who might benefit from the proposed model. We also posted flyers at the Clinics and invited potential participants to call Ms. Fuentes to find out more about the study and intervention.
Period: Overall Study
Arm/Group | Group Navigation Model
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Participants were Spanish-speaking Latinas with low income status living in the United States.
Arm/Group | Class
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Depression
Description: Patient Health Questionnaire-9 (PHQ-9) administered to monitor if intervention changes depression score. PHQ-9 total score for the nine items ranges from 0 to 27. Higher scores indicate increased depression. Scores of 5, 10, 15 and 20 represent cutpoints for mild, moderate, moderately severe and severe depression respectively.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Class
Number analyzed (Participants) | 21
score on a scale | 13.3 (5.8)

ADVERSE EVENTS:
Description: Adverse events were not monitored because this was a psychosocial study with minimal risks to participants.
Arm/Group | Class
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-03-30): https://cdn.clinicaltrials.gov/large-docs/30/NCT03901430/Prot_SAP_000.pdf
  • Informed Consent Form (2018-06-28): https://cdn.clinicaltrials.gov/large-docs/30/NCT03901430/ICF_001.pdf